CLINICAL TRIAL: NCT02778763
Title: Double Blind, Randomized, Placebo-controlled, Multicenter Pilot Study on Efficacy and Safety of CBLB612 Following Single Administration for Neutropenia Prophylaxis in Breast Cancer Patients Receiving Doxorubicin and Cyclophosphamide Myelosuppressive Chemotherapy
Brief Title: Study on Efficacy and Safety of CBLB612 for Neutropenia Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLab 612 LLC (Industry)
Collaborators: Cleveland BioLabs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BL-612-BC1
Record Dates: First submitted 2016-03-17; First posted 2016-05-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; TLR2; Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- One injection of CBLB612 after Сhemo (Experimental): One injection of placebo at Day -2 (48 hours prior AC chemotherapy treatment) and one injection of 4 μg CBLB612 at Day 1 (24 hours after AC chemotherapy treatment)
  Interventions: Drug: CBLB612; Drug: Placebo
- One injection of CBLB612 prior Сhemo (Experimental): One injection of 4 μg CBLB612 at Day -2 (48 hours prior AC chemotherapy treatment) and one injection of placebo at Day 1 (24 hours after AC chemotherapy treatment)
  Interventions: Drug: CBLB612; Drug: Placebo
- Placebo (Placebo Comparator): Two injections of placebo at Day -2 and Day 1 (48 hours prior and 24 hours after AC chemotherapy treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBLB612 — 4 μg CBLB612 SQ
  Arms: One injection of CBLB612 after Сhemo; One injection of CBLB612 prior Сhemo
Drug: Placebo
  Other Names: PBS; Phosphate buffer saline

SUMMARY:
Double blind, randomized, placebo-controlled, multicenter pilot study on efficacy and safety of CBLB612 following single administration for neutropenia prophylaxis in breast cancer patients receiving doxorubicin and cyclophosphamide myelosuppressive chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for the study participation.
2. Women in the age above 18 years inclusively.
3. Patients with histologically proven diagnosis of breast cancer to which the 1-st cycle of AC chemotherapy treatment is indicated (with 3-week interval).
4. ECOG Performance Status of 0-2.
5. Life expectancy ≥ 6 months.
6. Completion of all previous cancer therapies (including surgery, radiotherapy, chemotherapy, immunotherapy or study therapy) not later than 4 weeks prior the CBLB612 study.
7. All acute toxic effects of any previous therapies <Grade 1 prior the study, except for alopecia and/or neurotoxicity (Grade 1 or 2 is allowed).
8. Adequate hematopoiesis function:

   * WBC ≥3.0 x 103/μl;
   * PTT ≥1.5 x 103/μl;
   * Platelets ≥75 x 103/μl;
   * Hemoglobin ≥10 g/dl.
9. Adequate hepatic function:

   * Total bilirubin ≤1.5 x ULN;
   * ALT and AST ≤3 x ULN;
   * Alkaline phosphatase ≤2.5 x ULN.
10. Adequate renal function:

    * Creatinine ≤1.5 x ULN.
11. Adequate values of hemostasis system:

    * Prothrombin time;
    * ≤1.5 x ULN;
    * Activated partial thromboplastin time ≤1.5 x ULN;
    * INR ≤1.5 x ULN.
12. Adequate cardiac function which means

    * LVEF ≥45 based on ultrasonic examination of the heart or radionuclide angiography;
    * 12-lead electrocardiogram (ECG) with normal tracing, non-clinically significant changes may occur that do not require medical intervention.
13. Negative test for serological infection markers:

    * Negative HIV-antibody test;
    * Negative test for hepatitis B surface antigen (HBsAg);
    * Negative test for hepatitis C virus antibodies or negative test for mRNA of hepatitis C virus;
    * Negative test for Treponema pallidum antibodies.
14. Negative pregnancy test.
15. Consent of a patient with preserved reproductive function to use effective contraception method since screening up to at least 3 months after the study therapy.

    * e.g. intrauterine device, oral contraceptive, subcutaneous implant or double-barrier method (condom with contraceptive sponge or contraceptive vaginal suppository).
16. A patient shall be ready and able to meet the requirements of the study protocol and have the opportunity to participate in the study throughout the scheduled period.

Exclusion Criteria:

1. Rapidly progressing, clinically unstable breast cancer with present clinical signs of cerebral or meningeal membrane metastases.
2. Specific contraindications or hypersensitivity data in relation to any of the following drugs: doxorubicin, cyclophosphamide, CBLB612, anti-emetic agents (aprepitant, palonosetron), anti-inflammatory drugs (including paracetamol and aspirin), as well excipients of the abovementioned drug agents including polysorbate 80.
3. History of febrile neutropenia.
4. Presence of autoimmune disease.
5. Acute or chronic/relapsing inflammatory eye disease or any other significant eye disorder.

   * patients with mild and moderate myopia or hypermetropia, or presbyopia may be enrolled to the study.
6. Pregnancy or breast feeding, refusal to use adequate contraception methods during the study.
7. Signs of ongoing systemic bacterial, fungal or viral infectious disease or local infection requiring treatment at the randomization.

   * patients with local fungal lesion of skin area or nail may be enrolled to the study.
8. Systemic antibiotic therapy during up to 72 hours prior the randomization.
9. Previous radiotherapy of ≥30% of bone marrow.
10. Surgery or chemotherapy or experimental drug therapy within 4 weeks prior randomization.
11. Transplantation of bone marrow or peripheral blood precursor cells.
12. Intake of more than 10 portions of alcoholic beverages per week or anamnestic data on alcoholism, narcomania, drug abuse.

    * one portion of alcoholic beverage is 250 ml of beer, 125 ml of wine or 30 ml of strong alcoholic beverage.
13. Current immunosuppressant therapy including systemic corticosteroid therapy.
14. Clinically significant abnormal vital signs, results of laboratory and instrumental tests, based on the investigator assessment.
15. Any disease, condition, organ dysfunction or central nervous system disorder of the intake of narcotic drugs which, according to the investigator, may affect ability to participate in the study or hinder assessment of study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Duration of ANC <1.0 x 103/μl (Grade 3-4) | Baseline to up to 38 days after the 1st drug administration
Duration of ANC <0.5 x 103/μl (Grade 4) | Baseline to up to 38 days after the 1st drug administration
Maximum level of ANC decrease (nadir) | Baseline to up to 38 days after the 1st drug administration
Time to recovery of ANC level ≥1.5 x 103/μl | Baseline to up to 38 days after the 1st drug administration
Incidence of febrile neutropenia (simultaneous drop of ANC <0.5 x 103/μl and body temperature >38.0°C) | Baseline to up to 38 days after the 1st drug administration
Safety evaluation as measured by treatment-related adverse events as assessed by CTCAE v4.0 | Baseline to up to 38 days after the 1st drug administration

SECONDARY OUTCOMES:
Duration of thrombocytopenia <50 x 103/μl | Baseline to up to 38 days after the 1st drug administration
Duration of thrombocytopenia <25 x 103/μl | Baseline to up to 38 days after the 1st drug administration
Duration of thrombocytopenia <10 x 103/μl | Baseline to up to 38 days after the 1st drug administration
Maximum decrease of platelet level (nadir) | Baseline to up to 38 days after the 1st drug administration
Time to platelet level recovery ≥75 x 103/μl | Baseline to up to 38 days after the 1st drug administration
Changes in comparison with baseline level CD34+ by FACS | Baseline to up to 11 days after the 1st drug administration
Changes in comparison with baseline level absolute reticulocyte count | Baseline to up to 24 days after 1st the drug administration
Change of concentration of G-CSF by ELISA | Baseline to up to 11 days after the 1st drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A. Tiuliandin, MD PhD, Principal Investigator — Federal State Budgetary Institution "Russian Oncological Research Center named after N. N. Blokhin" of the Russian Academy of Medical Sciences; Aleksei G. Manikhas, MD PhD, Principal Investigator — St.-Petersburg State Budgetary Healtcare Institution "City Clinical Oncological Dispensary"; Dmitrii A. Krasnozhon, MD PhD, Principal Investigator — State Budgetary Healtcare Institution "Leningrad Region Oncological Dispensary"; Ruslan M. Paltuev, MD PhD, Principal Investigator — Non-State Healtcare Institution "Road Clinical Hospital of Open Joint Stock Company Russian Railways"; Natalia V. Fadeeva, MD PhD, Principal Investigator — Federal State Budgetary Healtcare Institution "Chelyabinsk Regional Clinical Oncological Dispensary"; Roman S. Ponomarev, MD PhD, Principal Investigator — State Region Budgetary Healtcare Institution "Murmansk Region Oncological Dispensary"

REFERENCES:
- See also: Related Info — http://www.cbiolabs.com/cblb612